CLINICAL TRIAL: NCT03521388
Title: Efficacy of a Stepped Internet-based Program for Prevention and Early Intervention of Depression in Adolescents
Brief Title: Internet-based Program for Prevention and Early Intervention of Adolescent Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Collaborators: Comisión Nacional de Investigación Científica y Tecnológica (Other Government); Millennium Institute for Research in Depression and Personality (MIDAP) (Unknown)
Responsible Party: Principal Investigator, Vania Martínez-Nahuel, Principal Investigator, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FONDECYT 1161696
Record Dates: First submitted 2018-04-17; First posted 2018-05-11 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Depressive Symptoms
Keywords: depression; adolescence; prevention; early intervention; internet-based
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention consists of an Internet-based program. The program will last 3 months, with subsequent monthly reinforcement sessions for other 3 months.
  The program is stepped, so that the more depressive symptomatology the more intensive program and consists of more components.
  The students will interact with the program via a monitoring and feedback e-mail with 3 questions of the PHQ--9- adolescent version (1st, 2nd & 9th question) that they will receive every 2 weeks and a Website that will allow them to access to psycho-educational videos and information. There will also in the Website sections that will provide emergency information, the possibility of a contact via e-mail, and group chats. Adolescents with more depressive symptoms or suicidal risk will be invited to participate in an online counselling appointment or a face to face assessment with a mental health professional of the program.
  Interventions: Behavioral: Take care of your mood (CUIDA TU ANIMO in Spanish)
- Control group (Other): The comparison group will receive general psychoeducation of depression in adolescents and will be on the waiting list to receive the intervention in the event that its efficacy is demonstrated.
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Take care of your mood (CUIDA TU ANIMO in Spanish) — The adolescents will be registered in the Website www.cuidatuanimo.org
  Arms: Intervention group
Other: Control — The adolescents will visit the Website www.cuidatuanimo.org, but they can not register
  Arms: Control group

SUMMARY:
Background: Depression is prevalent and can have devastating effects on the life of adolescents. Computerized intervention programs for depression have shown positive results. There is less evidence in prevention and early treatment for depression in Latin American adolescents.

Purpose: The purpose of this study is to determine whether a stepped internet-based program is effective to prevent and early intervene depression in adolescents attending 9th to 11th grade in eight schools in Santiago, Chile.

Study design: A two-arm cluster-randomized clinical trial will be carried out with approximately 600 adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Attending from ninth grade to eleventh grade in the eight participating schools.
* Informed consent and informed assent.
* Score in the depression questionnaire PHQ-9 adolescent version between 5 and 14.

Exclusion Criteria:

* High suicide risk defined by score in question 9 of the PHQ-9 adolescent version of 2 or more.
* Current treatment with antidepressant drugs.
* Current treatment with psychotherapy.

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 947 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Depressive Symptoms | 6 months after baseline assessment
  Patient Health Questionnaire-9 (PHQ-9) adolescent version, total score varies between 0 and 27, higher values represent a worse outcome

SECONDARY OUTCOMES:
Depressive Symptoms | 12 months after baseline assessment
  Patient Health Questionnaire-9 (PHQ-9) adolescent version, total score varies between 0 and 27, higher values represent a worse outcome
Anxiety Symptoms | 6 and 12 months after baseline assessment
  Generalized Anxiety Disorder-7 (GAD-7) adolescent version, total score varies between 0 and 21, higher values represent a worse outcome
Health-Related Quality of Life Index | 6 and 12 months after baseline assessment
  KIDSCREEN-10 index, total score varies between -3.53 and 83.8, higher values represent a better outcome
Social Problem Solving Skills | 6 and 12 months after baseline assessment
  Social Problem Solving Inventory-Revised Short Form (SPSI-RS), positive problem subscale orientation, and rational problem solving subscale, total score of each subscale varies between 0 to 20, higher scores represent better outcome
Dysfunctional Thoughts | 6 and 12 months after baseline assessment
  Children's Automatic Thought Questionnaire (CATS), personal failure subscale, total score of the subscale varies between 0 and 40, higher values represent worse outcome
Emotion Regulation | 6 and 12 months after baseline assessment
  Emotion Regulation Questionnaire (ERQ), reappraisal subscale, total score of the subscale varies between 6 and 42, higher values represent better outcome
Depression Stigma | 6 and 12 months after baseline assessment
  Depression Stigma Scale (DSS), personal stigma subscale, total score of the subscale varies between 0 and 36, higher values represent worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Vania Martinez, PhD, Principal Investigator — University of Chile
Locations (1):
- CEMERA, Faculty of Medicine, Universidad de Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No